CLINICAL TRIAL: NCT00205088
Title: The Use of Shunt Tap in Assessing Ventriculoperitoneal (VP) Shunt Malfunction
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2002-253
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-06

CONDITIONS: Signs or Symptoms of Shunt Failure

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The objective of the study is to test the sensitivity and specificity of a shunt tap to predict shunt failure.

ELIGIBILITY:
Inclusion Criteria:

* The patient has clinically suspected shunt malfunction.
* The patient has had an imaging study of the head.
* The patient needs a shunt revision.

Exclusion Criteria:

* The patient has not had an imaging study of the head.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bermans Iskandar, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States